CLINICAL TRIAL: NCT06921616
Title: A Multicenter, Randomized Controlled Clinical Trial on the Efficacy and Safety of Neuroendoscopic Hematoma Evacuation Combined With Methylprednisolone Sodium Succinate in the Treatment of Lobar Intracerebral Hemorrhage at the Early Stage.
Brief Title: Neuroendoscopic Hematoma Evacuation Combined With Methylprednisolone Sodium Succinate in the Treatment of Lobar Intracerebral Hemorrhage at the Early Stage.
Acronym: HEMS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yong Jiang (Other)
Responsible Party: Sponsor-Investigator, Yong Jiang, Prof., The Affiliated Hospital Of Southwest Medical University
Organization: The Affiliated Hospital Of Southwest Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025134
Record Dates: First submitted 2025-04-09; First posted 2025-04-10 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Intracerebral Hemorrhage Lobar; Methylprednisolone; Surgery
MeSH Terms: conditions — Stroke | interventions — Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The neuroendoscopic treatment group (Active Comparator): For patients with spontaneous lobar hemorrhage within 24 hours after the onset, simple neuroendoscopic hematoma evacuation was performed.
  Interventions: Procedure: Simple neuroendoscopic hematoma evacuation
- The methylprednisolone sodium succinate combined with neuroendoscopic treatment group (Experimental): For patients with spontaneous lobar hemorrhage within 24 hours after the onset, neuroendoscopic hematoma evacuation combined with methylprednisolone sodium succinate treatment was carried out.
  Interventions: Combination Product: Neuroendoscopic hematoma evacuation combined with sodium methylprednisolone succinate

INTERVENTIONS:
Procedure: Simple neuroendoscopic hematoma evacuation — For patients with spontaneous intracerebral hemorrhage within 24 hours after the onset of the disease, only simple neuroendoscopic evacuation of hematoma will be performed
  Arms: The neuroendoscopic treatment group
Combination Product: Neuroendoscopic hematoma evacuation combined with sodium methylprednisolone succinate — For patients with spontaneous intracerebral hemorrhage within 24 hours after the onset of the disease, they will be treated with the combination of neuroendoscopic hematoma evacuation and sodium methylprednisolone succinate.
  Administer sodium methylprednisolone succinate for injection by intravenous injection 6 hours after the onset of the disease. Specific administration: Intravenous injection at a dosage of 2 mg/kg, once daily, for three consecutive days.
  Arms: The methylprednisolone sodium succinate combined with neuroendoscopic treatment group

SUMMARY:
The aim of this trial is to investigate whether neuroendoscopic hematoma evacuation combined with early use of methylprednisolone sodium succinate can improve the efficacy and safety in the treatment with that of simple neuroendoscopic surgery alone for patients with spontaneous lobar intracerebral hemorrhage within 24 hours after the onset.

DETAILED DESCRIPTION:
There is still a lack of the best evidence-based reference for the treatment of lobar intracerebral hemorrhage. The ENRICH trial published in 2024 demonstrated that minimally invasive hematoma evacuation might have a better clinical prognosis than standard medical treatment in patients with spontaneous intracerebral hemorrhage. However, the significant effect of the surgery might be mainly attributed to the intervention in patients with lobar hemorrhage. Besides, simply relying on surgical removal of hematoma may not be sufficient to significantly improve the long-term prognosis of patients. How to effectively control secondary brain injury, reduce cerebral edema and inflammatory response is the key to improving the prognosis of patients with lobar intracerebral hemorrhage. Methylprednisolone sodium succinate can reduce the disruption of the blood-brain barrier and inflammatory response in animal models of intracerebral hemorrhage, and alleviate brain injury. The results of the MARVEL trial released in 2024 showed that methylprednisolone sodium succinate has demonstrated the potential to reduce the incidence of secondary intracerebral hemorrhage (ICH) and mortality in patients with acute ischemic stroke.

This study aims to systematically evaluate the efficacy and safety of neuroendoscopic hematoma evacuation combined with the early use of methylprednisolone sodium succinate in patients with lobar intracerebral hemorrhage through a multicenter, prospective, randomized controlled clinical trial. The study will compare the differences in main endpoint indicators such as functional independence, quality of life and survival rate at 3 months and 6 months after surgery between the group receiving surgical treatment combined with methylprednisolone sodium succinate and the group receiving surgical treatment alone, so as to explore the impact of different treatment strategies on the prognosis of patients with lobar intracerebral hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

1. The age ranges from 18 to 80 years old.
2. Diagnosed as spontaneous intracerebral hemorrhage (ICH) by cranial computed tomography (CT) examination, with the bleeding site located in the lobar region of the brain.
3. Calculate the hematoma volume according to the cranial CT examination, which should be within the range of 30 to 80 ml, and the shift of the midline structure at the level of the pineal gland is less than 3 mm. The formula for calculating the hematoma volume V (cubic centimeters) is V = A × B × C × 1/2. Here, A represents the longest diameter (in centimeters) of the largest hematoma layer on the horizontal position of the plain CT scan, B refers to the widest diameter (in centimeters) of the hematoma perpendicular to A on this plane, and C stands for the thickness (in centimeters) of the hematoma shown on the CT film.
4. The time interval from the onset of the disease to randomization is within 24 hours. In case the actual onset time is not clear, the onset time will be regarded as the time when the subject was last confirmed to be in good health.
5. The National Institutes of Health Stroke Scale (NIHSS) score ≥ 6 points at the time of randomization.
6. The Glasgow Coma Scale (GCS) score is between 5 and 14 points at the time of randomization.
7. The modified Rankin Scale (mRS) score is 0-1 points prior to the onset of the disease.
8. The patient and his or her legal representative sign the written informed consent form.

Exclusion Criteria:

1. Hemorrhage in other locations (e.g., hemorrhage in infratentorial sites such as the basal ganglia, thalamus, brainstem, or cerebellum).
2. Hemorrhage due to other causes (e.g., hemorrhage resulting from aneurysm, arteriovenous malformation, brain trauma, brain tumor, hemorrhagic transformation of large-area cerebral infarction, hemorrhage caused by amyloid angiopathy, hemorrhage due to coagulation disorders) or complicated by aneurysm, arteriovenous malformation, brain trauma, brain tumor, large-area cerebral infarction, amyloid angiopathy, severe coagulation disorders.
3. Patients with intraventricular hemorrhage or those in whom intracerebral hemorrhage (ICH) has ruptured into the ventricles and who are considered to require external ventricular drainage.
4. A history of any parenchymal brain hemorrhage or other intracranial subarachnoid, subdural, or epidural hemorrhage and a history of relevant surgeries within the past 30 days.
5. Patients with genetic or acquired bleeding tendencies, coagulation disorders such as deficiency of coagulation factors.
6. Platelet count < 75 × 10⁹/L.
7. Undergoing anticoagulant drug treatment with warfarin, dabigatran, or rivaroxaban, etc. within one week before enrollment, and having an international normalized ratio (INR) > 1.4.
8. Expected to require long-term anticoagulation and antiplatelet therapy.
9. A history of previous internal hemorrhage, with risks of gastrointestinal bleeding (such as gastrointestinal ulcers), genitourinary bleeding, or respiratory tract bleeding that has not been fully controlled.
10. Myocardial infarction occurring within the past 30 days.
11. Known to have a high embolism risk, including patients with mechanical heart valves implanted in vivo, a history of left heart thrombus, mitral stenosis accompanied by atrial fibrillation, acute pericarditis, or subacute bacterial endocarditis. Atrial fibrillation without mitral stenosis is eligible.
12. Severe liver function impairment, with alanine aminotransferase (ALT) > 3 times the upper limit of the normal range, or aspartate aminotransferase (AST) > 3 times the upper limit of the normal range. Severe renal insufficiency, with a glomerular filtration rate < 30 ml/min/1.73 m².
13. Patients with Alzheimer's disease or mental disorders who are unable to complete the follow-up plan as required.
14. Complicated by any severe diseases that, upon evaluation, may interfere with the trial results, including diseases of the respiratory system, circulatory system, digestive system, genitourinary system, endocrine system, immune system, and hematopoietic system, etc.
15. Allergic to drugs or devices related to the operation.
16. Pregnant or lactating women, or those planning to become pregnant within one year.
17. In the terminal stage of any disease with an expected lifespan of less than 6 months.
18. Currently participating in other clinical trials or having been previously enrolled in this trial.
19. The patient or his/her legal guardian is unwilling to sign the written informed consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin scale score (mRS) | 180 days
  disability level. The presence of impairments determines the transitions from mRS score 0 to mRS score 1 (symptoms) and mRS score 5 to mRS score 6 (death).
The mortality rate | 30 days
  evaluate death rate of the two treatment groups

SECONDARY OUTCOMES:
Proportion of patients non-disabled (Modified Rankin scale score (mRS) 0 to 1) | 180 days
  excellent outcome
Proportion of patients functionally independent (Modified Rankin scale score (mRS) 0 to 2) | 180 days
  functional independence
Proportion of patients ambulatory or bodily needs-capable or better (Modified Rankin scale score (mRS) 0 to 3) | 180 days
  ambulatory or bodily needs-capable or better
Change in National Institute of Health stroke scale (NIHSS) score between baseline and 7~10d or at discharge | 7~10 days or at discharge
  neurological changes. The scoring range is from 0 to 42 points. The higher the score is, the more severe the degree of neurological impairment in patients will be.
Change in Glasgow Coma Scale(GCS) between baseline and 7~10d or at discharge | 7~10 days or at discharge
  evaluate the state of consciousness. The scoring range is from 3 to 15 points. The lower the score is, the worse the patient's conscious state will be.
Improvement in residual hematoma volume between baseline and 7d or at discharge | 7~10 days or at discharge
Barthel Index Score(BI) | 180 days
  evaluate the Activities of Daily Living.The scoring range is from 0 to 100 points. The lower the score is, the poorer the patient's activities of daily living ability will be.
European Quality Five Dimensions Five Level scale (EQ-5D-5L) | 180 days
  Health-related quality of life. The scoring range is from 5 to 25 points. The higher the score is, the poorer the patient's health-related quality of life will be.
Mortality within 7 days randomly or at discharge | 7days or at discharge
  evaluate death rate of the two treatment groups
symptomatic intracranial rebleeding, asymptomatic intracranial rebleeding and intracranial infection | within 30 days after randomized
symptomatic intracranial rebleeding, asymptomatic intracranial rebleeding and intracranial infection | within 180 days after randomized
severe adverse events | within 180 days after randomization
  evaluate complications and any adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Southwest Medical University, Luzhou, China, China

IPD SHARING:
Plan to Share IPD: No